CLINICAL TRIAL: NCT05814770
Title: Compare the Efficacy and Safety of Finerenone, a New Type of Mineralocorticoid Receptor Antagonist, and Spironolactone in the Treatment of Primary Aldosteronism: a Single-Center, Prospective, Randomized Controlled Study
Brief Title: Comparing the Efficacy and Safety of Finerenone and Spironolactone in the Treatment of Primary Aldosteronism
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: National Key Research and Development Program of China (Unknown); National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PA2023
Record Dates: First submitted 2023-03-13; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Primary Aldosteronism; Hypertension
Keywords: primary aldosteronism; hypertension; finerenone; spironolactone; treatment
MeSH Terms: conditions — Hyperaldosteronism; Hypertension | interventions — finerenone; Spironolactone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Finerenone (Experimental)
  Interventions: Drug: Finerenone
- Spironolactone (Active Comparator)
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Drug: Finerenone — The participants were randomized in an equal ratio to receive finerenone 10 mg once daily. Patients received the initial dose of study drug for the first 4 weeks of randomized treatment period. Thereafter, the dose of study medication was not changed for patients with adequate BP control. For patients not meeting BP < 140/90 mmHg at week 4, the dose of study medication was increased to finerenone 20 mg once daily. If BP > 160/110 mmHg at the time of 8 weeks follow-up, nifedipine 30mg once day was added.
  Other Names: Kerendia
  Arms: Finerenone
Drug: Spironolactone — The participants were randomized in an equal ratio to receive spironolactone 20 mg twice daily. Patients received the initial dose of study drug for the first 4 weeks of randomized treatment period. Thereafter, the dose of study medication was not changed for patients with adequate BP control. For patients not meeting BP < 140/90 mmHg at week 4, the dose of study medication was increased to spironolactone 40 mg twice daily. If BP > 160/110 mmHg at the time of 8 weeks follow-up, nifedipine 30mg once day was added.
  Arms: Spironolactone

SUMMARY:
Primary aldosteronism (PA) is thought to be the most common secondary endocrine form of hypertension. Compared with patients with essential hypertension with similar blood pressure, patients with PA have significantly higher atrial fibrillation, myocardial infarction, heart failure, stroke, deterioration of renal function and all-cause mortality. Therefore, early and systematic implementation of effective surgical or medical treatment is essential to prevent or reverse the excess vascular events and mortality of these patients. The patients with bilateral PA were mainly treated with mineralocorticoid receptor antagonists (MRAs). The MRA spironolactone is effective at lowering BP and reversing the harmful metabolic consequences, but its use is limited by adverse effects such as gynaecomastia, mastodynia, menstrual abnormalities and impotence due to its agonist activity at the progesterone receptor and antagonist activity at the androgen receptor. Finerenone is claimed to be a more selective blocker of the mineralocorticoid receptor than spironolactone being associated with fewer antiandrogenic side-effects. In this study, we will compare the efficacy, safety and tolerability of finerenone versus spironolactone in patients with hypertension associated with primary aldosteronism.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age: 18-75 years old.
* 2.History of hypertension, DBP <120 mmHg, SBP <180 mmHg.
* 3.Serum potassium level ≥ 2.5 mmol/L.
* 4.Primary Aldosteronis diagnosed by increased aldosterone renin ratio (ARR) > 30 ng/dl: ng/ml/h, and serum aldosterone levels ≥15 ng / dl, and confirmed by captopril inhibition test.

Exclusion Criteria:

* 1. Abnormal renal function: serum creatinine ≥ 2 × ULN or eGFR ≤ 60 ml/(min * 1.73m2);
* 2. Abnormal liver function: ALT and AST ≤ 2.5 × ULN, TBIL ≤ 1.5 × ULN；
* 3. Cardiac insufficiency, acute myocardial infarction, stroke or other acute cardiovascular events within 6 months;
* 4. Take spironolactone, guanethidine or reserpine 30 days before enrollment;
* 5. Known or suspected tumor; Other autoimmune diseases, uncontrolled infectious diseases, serious respiratory, blood and nervous system diseases;
* 6. There is a pregnancy plan in pregnancy or 3 months before and after treatment. Breast-feeding women;
* 7. Those who have mental illness, alcohol or drug abuse and cannot cooperate with treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Hypertension remission rate. | 12 weeks.
  The proportion of patients with blood pressure<140/90 mmHg at 12 weeks.

SECONDARY OUTCOMES:
The change of systolic and diastolic BP from the baseline level. | Baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks.
  To compare the antihypertensive effect of finerenone versus spironolactone and to establish the noninferiority of finerenone by measuring the mean change from baseline to the week 16 endpoint in end- of-dose (trough) seated DBP.
Change of serum potassium level | Baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks.
  Change of serum potassium level (mmol/L)
Changes of plasma renin activity and ARR. | Baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks.
Incidence of Treatment-Adverse Events as assessed by gynaecomastia, mastodynia, menstrual abnormalities, impotence, hyperkalemia and other adverse events. | Baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks.
  1. Adverse effects such as gynaecomastia, mastodynia, menstrual abnormalities and impotence due to its agonist activity.
  2. Hyperkalemia.
  3. Other adverse events.
Proportion of patients with normal serum. | Baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Li, Study Director — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School